CLINICAL TRIAL: NCT06074172
Title: The Effect of Cannabidiol in Learning and Memory of Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: Institute of Cannabis Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MD012420BM
Record Dates: First submitted 2023-09-26; First posted 2023-10-10 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Memory
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Two-arm Case-Crossover
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple (Participant, Care Provider, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo, Then Cannabidiol (Placebo Comparator): Participants first received a Placebo 246 mg press pill during visit 1. After a washout period of 1 week, subjects received a Cannabidiol press pill during visit 2.
  Interventions: Drug: Placebo (246mg press pill)
- Cannabidiol, Then Placebo (Active Comparator): Participants first received a Cannabidiol 246 mg press pill during visit 1. After a washout period of 1 week, subjects received a Placebo press pill during visit 2.
  Interventions: Drug: Cannabidiol (246mg press pill)

INTERVENTIONS:
Drug: Cannabidiol (246mg press pill) — Cannabidiol press pills provided by Steve Goods CBD (Longmont, Colorado). CBD pills were tested by the chemistry lab at CSU Pueblo and by Botanacor in Denver, CO. Both laboratories determined CBD pills to be 99.98% pure with no THC, heavy metals, bacteria, and pesticides detected.
  Arms: Cannabidiol, Then Placebo
Drug: Placebo (246mg press pill) — Placebo press pills were provided by Steve Goods CBD (Longmont, Colorado). Placebo pills were tested by the chemistry lab at CSU Pueblo and by Botanacar in Denver, CO. Both laboratories determined placebo pills to be pure with no heavy metals, bacteria, and pesticides detected.
  Arms: Placebo, Then Cannabidiol

SUMMARY:
The main objectives of this study were to test if a singular dose of Cannabidiol (1) enhances the learning and memory of healthy human subjects, (2) test if Cannabidiol has negative effects on Retroactive and Proactive Interference during learning, (3) and test if demographic factors will influence CBD's modulation of human learning and memory.

DETAILED DESCRIPTION:
Using a randomized, double-blind, placebo-controlled two-arm case-crossover trial, this study investigates the effect of 246 milligrams (mg) of Cannabidiol (CBD) on the learning and memory scores of human subjects, as well as the effect of Cannabidiol on Proactive and Retroactive Interference. This study also investigated the influence of demographic factors on CBD's modulation of human learning and memory.

This study was conducted at Colorado State University-Pueblo (CSU Pueblo) with volunteers recruited from CSU Pueblo and the local Pueblo community. Fifty-seven subjects were randomized in a double-blind manner to receive either CBD or placebo before completing two versions of learning and memory assessments. Each version of the learning and memory assessment included the Montreal Cognitive Assessment (MOCA), the Rey Auditory Verbal Learning Task-Revised (RAVLT-R), and the Logical Memory Subject of the Weschler Memory Scale. Several components of the RAVLT-R were evaluated including the Sum of Trials (Trials I-V) score, Proactive Interference Ratio (PI Ratio), and Retroactive Interference (RI Ratio).

ELIGIBILITY:
Inclusion Criteria:

* Were 18 years of age or older

Exclusion Criteria:

* Were pregnant or breast-feeding
* Had been diagnosed with mental illness
* Didn't speak English fluently
* Had severe hearing problems
* Had recreational or opioid drug contaminants in their urine
* Were involved in criminal activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-03-14 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moussa M Diawara, PhD, Principal Investigator — Colorado State University-Pueblo
Locations (1):
- Colorado State University Pueblo, Pueblo, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual (de-identified) participant data is to be made available to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available upon request.
Access Criteria: Data will become available upon request.

REFERENCES:
- [Derived] Gebregzi HH, Zeiger JS, Smith JP, Stuyt L, Cullen L, Carsella J, Rogers DC, Lafebre J, Knalfec J, Vargas A, Diawara MM. Oral cannabidiol did not impair learning and memory in healthy adults. J Cannabis Res. 2025 Jan 23;7(1):5. doi: 10.1186/s42238-025-00262-2. PMID 39849639

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Visit 1 Drug Administration): 246mg Placebo, oral, single-dose (visit 1 drug administration)
  Placebo in Oral Dose Form: Placebo press pills provided by Steve Goods CBD (Longmont, Colorado). Placebo pills were tested by the chemistry lab at CSU Pueblo and by Botanacar in Denver, CO. Both laboratories determined placebo pills to be pure with no heavy metals, bacteria, and pesticides detected.
- Cannabidiol (Visit 1 Drug Administration): 246mg Cannabidiol, oral single-dose (visit 1 drug administration)
  Cannabidiol in Oral Dose Form: Cannabidiol press pills provided by Steve Goods CBD (Longmont, Colorado). CBD pills were tested by the chemistry lab at CSU Pueblo and by Botanacor in Denver, CO. Both laboratories determined CBD pills to be 99.98% pure with no THC, heavy metals, bacteria, and pesticides detected.
Period: Overall Study
Arm/Group | Placebo (Visit 1 Drug Administration) | Cannabidiol (Visit 1 Drug Administration)
Started | 27 | 30
Completed | 21 | 23
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Population: Enrollment was stopped after interim analyses were completed. 57 subjects were enrolled in the study, but 35 were included in the final analyses. Subjects were required to come for visits 1 and 2. A large dropout between visits 1 and 2 was due to the COVID pandemic which caused for subjects to be lost to follow up. The baseline characteristics are reported for the 35 repeat subjects which is representative of the participant population that results were reported for.
Groups:
- Placebo First, Then Cannabidiol: 246mg Placebo, oral, single-dose (visit 1 or visit 2 drug administration)
  Placebo in Oral Dose Form: Placebo press pills provided by Steve Goods CBD (Longmont, Colorado). Placebo pills were tested by the chemistry lab at CSU Pueblo and by Botanacar in Denver, CO. Both laboratories determined placebo pills to be pure with no heavy metals, bacteria, and pesticides detected.
- Cannabidiol First, Then Placebo: 246mg Cannabidiol, oral single-dose (visit 1 or visit 2 drug administration)
  Cannabidiol in Oral Dose Form: Cannabidiol press pills provided by Steve Goods CBD (Longmont, Colorado). CBD pills were tested by the chemistry lab at CSU Pueblo and by Botanacor in Denver, CO. Both laboratories determined CBD pills to be 99.98% pure with no THC, heavy metals, bacteria, and pesticides detected.
- Total: Total of all reporting groups
Arm/Group | Placebo First, Then Cannabidiol | Cannabidiol First, Then Placebo | Total
Number analyzed (Participants) | 16 | 19 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 19 | 35
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 27 [19 to 64] | 33 [18 to 63] | 30 [18 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 9 | 14
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 12 | 10 | 22
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 19 | 35
History of CBD Use, categorical [Count of Participants; unit: Participants]
  Non-user | 12 | 16 | 28
  User | 4 | 3 | 7
Urine THC Result, categorical [Count of Participants; unit: Participants]
  THC - | 7 | 12 | 19
  THC + | 9 | 7 | 16
History of Nicotine Use, categorical [Count of Participants; unit: Participants]
  Non-user | 14 | 15 | 29
  User | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Sum of Trials (I-V)
Description: Sum of Trials = Trial A1 + Trial A2 + Trial A3 + Trial A4 + Trial A5;
  Trial A1/A2/A3/A4/A5 are in reference to each trial in which list A is recalled during memory encoding. The score range for Sum of Trials is 0 to 75. A higher score is indicative of greater performance on the memory test and a lower score is indicative of lower performance on the memory test.
  Participants were instructed to listen to a list of 15 words (List A) read to them. Subjects were asked recall List A during five different trials (A1, A2, A3, A4, A5), with the words repeated to them after each trial. Participants were scored for the number of correctly repeated words for each trial.
Time Frame: Each trial is 45 seconds for encoding and recall
Population: The data reported is for 35 adult healthy human subjects who came in for visits 1 and 2 and were randomized to a treatment group (CBD or placebo). Since the 35 subjects came in twice, each of them received both interventions (CBD and placebo).
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Placebo (Administered During Visits 1 or 2): 246mg Placebo, oral, single-dose (visit 1 drug administration)
  Placebo in Oral Dose Form: Placebo press pills provided by Steve Goods CBD (Longmont, Colorado). Placebo pills were tested by the chemistry lab at CSU Pueblo and by Botanacar in Denver, CO. Both laboratories determined placebo pills to be pure with no heavy metals, bacteria, and pesticides detected.
- Cannabidiol (Administered During Visits 1 or 2): 246mg Cannabidiol, oral single-dose (visit 1 drug administration)
  Cannabidiol in Oral Dose Form: Cannabidiol press pills provided by Steve Goods CBD (Longmont, Colorado). CBD pills were tested by the chemistry lab at CSU Pueblo and by Botanacor in Denver, CO. Both laboratories determined CBD pills to be 99.98% pure with no THC, heavy metals, bacteria, and pesticides detected.
Arm/Group | Placebo (Administered During Visits 1 or 2) | Cannabidiol (Administered During Visits 1 or 2)
Number analyzed (Participants) | 35 | 35
score on a scale | 49.09 (1.85) | 47.17 (1.85)

2. Primary Outcome: Proactive Interference Ratio (PI Ratio)
Description: PI Ratio = Trial B1/A1. Proactive interference is the tendency for previously learned information to affect to hinder learning of new information. A higher proactive interference ratio indicates protective effects on memory i.e. protection from interference during learning. A lower proactive interference is indicative of negative effects on memory caused from interference. Trial A1 is in reference to list A recall during the first trial. Trial B1 is in reference to list B recall. Highest score for each trial is 15 with a point awarded for each correctly recalled word from List A (15 words) and List B (15 words).
Time Frame: Each trial is 45 seconds for encoding and recall
Population: Adult healthy human subjects
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Placebo (Visit 1 Drug Administration) | Cannabidiol (Visit 1 Drug Administration)
Number analyzed (Participants) | 35 | 35
ratio | 1.04 (0.08) | 1.21 (0.08)
Statistical Analysis 1: Comparison: Placebo (Visit 1 Drug Administration) vs Cannabidiol (Visit 1 Drug Administration); Test type: Other — Linear Mixed Models were done with a compound symmetry covariance structure. This infers that the variances (pooled within-group) and covariances (across subjects) of all of the repeated measures are homogenous; p = 0.008, Linear Mixed Model — In the Bonferroni corrected Linear Mixed Model for PI Ratio, the p-value for the following interaction was reported: Treatment*Age; Linear Mixed Model analyses: 1. Factor: Treatment group 2. Covariates: Age, Sex, CBD Use history, and Urine THC 3. Interactions

3. Primary Outcome: Retroactive Interference Ratio (RI Ratio)
Description: RI Ratio = Trial A6/A5. Retroactive interference is the tendency for newly learned information to hinder the memory of previously learned information. A higher retroactive interference ratio indicates protection from interference during learning. A lower retroactive interference ratio is indicative of negative effects on memory caused from interference. Trial A6 is referring to delayed recall of list A; Trial A5 is referring to the fifth trial of list A recall. Highest score for each trial is 15 with a point awarded for each word correctly recalled from List A (15 words).
Time Frame: Each trial is 45 seconds for encoding and recall
Population: Adult healthy human subjects
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Placebo (Visit 1 Drug Administration) | Cannabidiol (Visit 1 Drug Administration)
Number analyzed (Participants) | 35 | 35
ratio | 0.87 (0.03) | 0.83 (0.03)

4. Primary Outcome: Total Prose Recall
Description: Total Prose Recall = Immediate Recall + Delayed Recall; Recall of a prose story was done immediately then after a delay; Highest score for prose recall test is 25 with a point awarded for each item correctly recalled in the story (25 total items). A higher recall score is indicative of better memory.
Time Frame: Each recall takes about 5 min for encoding and recall
Population: Adult healthy human subjects
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo (Visit 1 Drug Administration) | Cannabidiol (Visit 1 Drug Administration)
Number analyzed (Participants) | 35 | 35
Score on a scale | 27.49 (1.46) | 25.49 (1.46)

5. Primary Outcome: Montreal Cognitive Assessment Score
Description: Assessment of basal cognitive function; The range for Montreal Cognitive Assessment (MOCA) scores is 0 to 30. A higher recall score is indicative of better performance on the memory test. A lower recall score is indicative of worse performance on the memory test.
Time Frame: 10 minutes total for encoding and recall
Population: Adult healthy human population
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo (Visit 1 Drug Administration) | Cannabidiol (Visit 1 Drug Administration)
Number analyzed (Participants) | 35 | 35
Score on a scale | 26.31 (0.46) | 26.63 (0.46)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected as subjects completed exit surveys at the end of visit 2. Completion of the exit survey took about 15-20 minutes. Assessment administrators also followed up with study participants up until the completion of the study to confirm whether any adverse events occurred or resolved. Study participants confirmed that all adverse events were resolved. Adverse event data was collected at the end of visit 2.
Description: An adverse event (AE) is an untoward medical occurrence in a patient who was administered an investigational product.
  A serious adverse event is an AE which also fulfills the following criteria:
  1. Results in death
  2. Is life-threatening
  3. Requires in-patient hospitalization
  4. Results in persistent or significant disability/incapacity
  5. Cause congenital anomaly/birth defect
  6. Important medical event that requires intervention to prevent permanent impairment or damage
Arm/Group | Placebo (Administered During Visits 1 or 2) | Cannabidiol (Administered During Visits 1 or 2)
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 1/35 | 4/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Administered During Visits 1 or 2) (N=35) | Cannabidiol (Administered During Visits 1 or 2) (N=35)
Drowsiness (Nervous system disorders) | 0 (0) | 4 (4) — Subjects were asked to complete an exit survey with possible adverse events or asked to fill in the line. 4 subjects reported drowsiness or fatigues.
Hunger (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participants were given an exit survey with a list of possible adverse events or asked to fill in the line. 1 Subject reported hunger.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-28): https://cdn.clinicaltrials.gov/large-docs/72/NCT06074172/Prot_SAP_002.pdf